CLINICAL TRIAL: NCT03485625
Title: Adjuncts to Intravenous Regional Anaesthesia, a Comparison Between Ketorolac and Paracetamol
Brief Title: Adjuncts to IVRA, a Comparison Between Ketorolac and Paracetamol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Rabiee Ali, Resident doctor at the department of anaesthesiology and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bier's block
Record Dates: First submitted 2018-03-21; First posted 2018-04-02 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Ketorolac; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine (Experimental): Patients in group C will receive 3 mg/kg of lidocaine 2% diluted with saline to a total volume of 40 ml.
  Interventions: Drug: Lidocaine
- Lidocaine+ Ketorolac (Experimental): Patients in group K receive 3 mg/kg of lidocaine 2% + 20 mg ketorolac diluted with saline to a total volume of 40 ml.
  Interventions: Drug: Lidocaine; Drug: Ketorolac
- Lidocaine+Paracetamol (Experimental): Patients in group P will receive 3 mg/kg of lidocaine 2% + 300 mg paracetamol diluted with saline to a total volume of 40 ml.
  Interventions: Drug: Lidocaine; Drug: paracetamol

INTERVENTIONS:
Drug: Lidocaine — Two cannulae were placed, one in a vein on the dorsum of the operative hand and the other on the non operative hand for i.v fluids. The operative arm was elevated for 2 min and was then exsanguinated with an elastic bandage. A pneumatic tourniquet was then placed around the upper arm, and the cuff was inflated to 100 mm Hg above systolic BP. Circulatory isolation of the arm was verified by inspection, absence of a radial pulse, and a loss of the pulse oximetry tracing in the ipsilateral index fingers The solutions were prepared by an anesthesiology assistant not involved in any part of the study. The solutions were injected over 90 s by an anaesthesiologist.
Drug: Ketorolac — Two cannulae were placed, one in a vein on the dorsum of the operative hand and the other on the non operative hand for i.v fluids. The operative arm was elevated for 2 min and was then exsanguinated with an elastic bandage. A pneumatic tourniquet was then placed around the upper arm, and the cuff was inflated to 100 mm Hg above systolic BP. Circulatory isolation of the arm was verified by inspection, absence of a radial pulse, and a loss of the pulse oximetry tracing in the ipsilateral index fingers The solutions were prepared by an anesthesiology assistant not involved in any part of the study. The solutions were injected over 90 s by an anaesthesiologist.
  Arms: Lidocaine+ Ketorolac
Drug: paracetamol — Two cannulae were placed, one in a vein on the dorsum of the operative hand and the other on the non operative hand for i.v fluids. The operative arm was elevated for 2 min and was then exsanguinated with an elastic bandage. A pneumatic tourniquet was then placed around the upper arm, and the cuff was inflated to 100 mm Hg above systolic BP. Circulatory isolation of the arm was verified by inspection, absence of a radial pulse, and a loss of the pulse oximetry tracing in the ipsilateral index fingers The solutions were prepared by an anesthesiology assistant not involved in any part of the study. The solutions were injected over 90 s by an anaesthesiologist.
  Arms: Lidocaine+Paracetamol

SUMMARY:
The study was planned to compare the effect of ketorolac 20 mg to 300 mg of paracetamol when added to lidocaine 3 mg/kg for Intravenous regional anaesthesia.

DETAILED DESCRIPTION:
All patients were premedicated 15 minutes before the surgical procedure with I.V. 0.06mg/kg of midazolam. In the operating room, patients were monitored for non invasive blood pressure (NIBP), oxygen saturation (Spo2) and pulse rate (PR).

Two cannulae were placed, one in a vein on the dorsum of the operative hand and the other on the non operative hand for i.v fluids. The operative arm was elevated for 2 min and was then exsanguinated with an elastic bandage. A pneumatic tourniquet was then placed around the upper arm, and the cuff was inflated to 100 mm Hg above systolic BP. Circulatory isolation of the arm was verified by inspection, absence of a radial pulse, and a loss of the pulse oximetry tracing in the ipsilateral index fingers. The solutions were prepared by an anesthesiology assistant not involved in any part of the study. The solutions were injected over 90 s by an anaesthesiologist. During surgery if patient reported pain during operation (VAS 4 or greater) inj. fentanyl 1 μg/kg was given and total amount used was recorded. Postoperatively patients were questioned for pain and if VAS > 4, 75 mg intramuscular diclofenac was given.Total amount used was recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status I or II, who will be scheduled for surgery of the hand or the forearm were included in this study after informed consent

Exclusion Criteria:

* Severe Raynaud's Disease
* Sickle Cell Disease
* Crush injury to the limb
* A history of allergic reaction to lidocaine
* Liver disease or kidney disease
* Significant cardiovascular disease
* Highly nervous and uncooperative patients
* Patient with history of opioid dependence
* Drug or alcohol abuse
* Psychiatric disorder
* Neurological diseases

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
The time to first analgesic request. | 1 year
  The time from tourniquet release until first patient request for analgesic

SECONDARY OUTCOMES:
sensory block | 1 year
  Onset of sensory block will be assessed by a pin prick performed at 1 minute interval in the dermatomal sensory distribution of the medial and lateral ante brachial cutaneous, ulnar, median and radial nerves. Sensory block onset time will be recorded as time elapsed from injection of drug to sensory block achieved in all dermatomes
motor block | 1 year
  Onset of motor block will be assessed by asking the subject to flex and extend his/her wrist and fingers.Complete motor block will be recorded when no voluntary movement will be possible.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Abdel-Baki Abdel-Rahman, Lecturer of anaesthesia, Study Chair — Assiut University
Locations (1):
- Omar Ali, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided